CLINICAL TRIAL: NCT03348722
Title: START (Active Surveillance or Radical Treatment for Newly Diagnosed Patients With a Localized, Low Risk, Prostate Cancer): an Epidemiological Study of the Oncology Network of Piemonte and Valle d'Aosta (Italy)
Brief Title: Active Surveillance or Radical Treatment for Newly Diagnosed Patients With a Localized, Low Risk, Prostate Cancer START
Acronym: START
Status: Completed | Type: Observational
Sponsor: Rete Oncologica Piemonte, Valle d'Aosta (Other)
Collaborators: Compagnia di San Paolo (Other); A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: START
Record Dates: First submitted 2017-06-19; First posted 2017-11-21 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Prostatic Neoplasm
Keywords: Active surveillance; Low risk prostate cancer; Prostatic neoplasm/therapy (MESH); Prostatic neoplasm/surgery (MESH); Prostatic neoplasm/radiotherapy (MESH); Prostatectomy (MESH); Quality of life (MESH); Costs and Cost Analysis (MESH)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Active surveillance: Newly diagnosed low risk prostate cancer patients managed according to an active surveillance program
  Interventions: Other: Active surveillance
- Radical prostatectomy: Newly diagnosed low risk prostate cancer patients undergoing radical prostatectomy
  Interventions: Procedure: Radical prostatectomy
- Radiotherapy: Newly diagnosed low risk prostate cancer patients undergoing radiotherapy (external or brachitherapy)
  Interventions: Radiation: Radiotherapy
- Other radical treatment: Newly diagnosed low risk prostate cancer patients undergoing other radical treatments (HIFU, cryotherapy, others)
  Interventions: Procedure: Other radical treatments

INTERVENTIONS:
Other: Active surveillance — PSA testing (every 3 months, then every 6 after 30 months), clinical visit and DRE every 6 months, prostate biopsy after 1, 4 and 7 years
  Groups: Active surveillance
Procedure: Radical prostatectomy — Radical prostatectomy (open, laparoscopic or robotic)
  Groups: Radical prostatectomy
Radiation: Radiotherapy — External radical radiotherapy or brachitherapy
  Groups: Radiotherapy
Procedure: Other radical treatments — High intensity focal ultrasound, cryotherapy, others
  Groups: Other radical treatment

SUMMARY:
The purpose of the START project is to evaluate the acceptability, the safety and the cost-effectiveness of a population based program of active surveillance for patients newly diagnosed with a localized, low risk, prostate cancer.

DETAILED DESCRIPTION:
Comparative effectiveness research project. All newly diagnosed prostate cancer patients fulfilling the low risk definition, resident in Piedmont or in Valle D'Aosta regions, will be invited to participate. All enrolled patients will receive full and clear information about their prognosis together with a balanced synthesis of the benefits and risks of the available treatments (active surveillance or radical treatments).

Specific objectives are:

* To estimate, at a population level, the proportion of newly diagnosed prostate cancer at low risk, eligible for active surveillance, the proportion of those accepting to be enrolled in a cohort of active surveillance and the risk of abandoning the program during follow-up.
* To compare the patients' and physicians' characteristics of those accepting to be managed within the active surveillance program with those preferring a radical treatment (either surgery or radiotherapy).
* To compare, at a population level, the clinical outcomes, quality of life and costs associated to different treatment choices.

ELIGIBILITY:
IInclusion Criteria:

1. Newly diagnosed low risk prostate cancer patients, defined according to the presence of all the following criteria:

   * diagnosis of adenocarcinoma of the prostate
   * prostate cancer clinical stage T1c o T2a
   * PSA <=10ng/ml at diagnosis
   * adequate biopsy sampling according to prostate volume
   * maximum of two positive cores for random sampling and of maximum two lesions for target biopsies (even if the number of positive samples if >2)
   * Gleason grade 3+3 ( in patients age>70 Gleason 3+4)
2. Residence in Piemonte or Valle D'Aosta regions;
3. Patients suitable for radical treatment (surgery or radiotherapy);
4. Age at diagnosis <= 75 years or >75 years if fragility assessment (measured with the G8 score)> = 14;
5. Patients suitability for expressing a valid consent to participate in the study.

Exclusion Criteria:

1. Patients previously treated for prostate cancer.
2. Patients not willing to undergo radical treatments (surgery or radiotherapy).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed low risk prostate cancer patients resident in Piemonte or in Valle D'Aosta regions (Northern Italy)
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Treatment-Free Survival (TFS) | Up to 24 months
  Proportion of patients in active surveillance program alive and not undergoing active treatment for prostate cancer.

SECONDARY OUTCOMES:
Quality of Life | Up to 24 months
  Measured through validated questionnaire EORTC QLQ-C30 at baseline and every six months during the first 2 years.
Quality of Life | Up to 24 months
  Measured through validated questionnaire QLQ-PR25 at baseline and every six months during the first 2 years.
Quality of Life | Up to 24 months
  Measured through validated questionnaire IPSS at baseline and every six months during the first 2 years.
Quality of Life | Up to 24 months
  Measured through validated questionnaire IIEF-5 at baseline and every six months during the first 2 years.
Quality of Life | Up to 24 months
  Measured through validated questionnaire HADS at baseline and every six months during the first 2 years.
Quality of Life | Up to 24 months
  Measured through validated questionnaire EuroQol-5D at baseline and every six months during the first 2 years.
Quality of Life | Up to 24 months
  Measured through validated questionnaire MHLC -Form C at baseline and every six months during the first 2 years.
Cost-effectiveness | Up to 24 months
  Incremental cost-effectiveness ratio calculated as the ratio between difference in costs and difference in QALYs (Quality Adjusted Life Years, from EQ-5D) among the treatment groups, during the first 2 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Bertetto, MD, Principal Investigator — Oncology Network of Piedmont and Valle d'Aosta
Locations (1):
- Oncolgy Network of Piemonte and Valle d'Aosta - Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: https://start.epiclin.it/home — https://start.epiclin.it/home